CLINICAL TRIAL: NCT06750991
Title: A Prospective, Open-label Phase II Study of Chidamide, Decitabine Plus R-CHOP in Previously Untreated Diffuse Large B-cell Lymphoma With a Combination of TP53 Mutation and Del(17p)
Brief Title: CD-RCHOP in ND DLBCL With a Combination of TP53 Mutation and Del(17p)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-B45
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: DLBCL
Keywords: DLBCL; TP53; Chidamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDR-CHOP (Experimental): Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of R-CHOP, followed by the remaining 5 cycles courses of chidamide and decitabine combined with a standard-dose R-CHOP regimen.
  Interventions: Drug: CDR-CHOP

INTERVENTIONS:
Drug: CDR-CHOP — Rituximab 375 mg/m2 D1 Cyclophosphamide 750 mg/m2 D2 Doxorubicin 50 mg/m2 D2 Vincristine 1.4 mg/m2 D2 Prednisone 69 mg.m2 D2-6 Chidamide 20 mg/d D1,4,8,11 Decitabine 10 mg/m2 D-5 - -1

SUMMARY:
This was an open, multicenter clinical study of newly treated DLBCL patients with TP53 mutations and del(17p) with IPI>1. Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of R-CHOP, followed by the remaining 5 cycles courses of chidamide and decitabine combined with a standard-dose R-CHOP regimen.

DETAILED DESCRIPTION:
This was an open, multicenter clinical study of newly treated DLBCL patients with TP53 mutations and del(17p) with IPI>1. Participants who met the inclusion/exclusion criteria signed informed consent and received 1 course of R-CHOP, followed by the remaining 5 cycles courses of chidamide and decitabine combined with a standard-dose R-CHOP regimen. . Patients who achieve CR will continue with chidamide maintenance therapy (20mg, D1,4,8,11) or opt for autologous hematopoietic stem cell transplantation after completion of induction therapy, with maintenance therapy recommended for at least 1 year (unless intolerable side effects or disease progression occur). Concurrent follow-up assessment (patients will enter the follow-up period described in the time and event table) until the end of the specified follow-up period (total study duration is 3 years) or until the patient meets the exit criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed diffuse large B-cell lymphoma with CD20 positive;
* 2. Pathologically confirmed a combination of TP53 mutation and del(17p);
* 3. Age ≥ 18 years old, ≦75 years old;
* 4. ECOG physical status score of 0, 1 or 2;
* 5. No previous history of malignant tumors; No other tumors occurred simultaneously;
* 6. Patients judged by the investigator to have a life expectancy of at least 6 months;
* 7. The patient or his legal representative must provide written informed consent prior to any research special examination or procedure.
* 8. International prognostic Index (IPI) >1 score.

Exclusion Criteria:

* 1. Have previously received systemic or local treatment including chemotherapy;
* 2. Previously received autologous stem cell transplantation;
* 3. Previous history of other malignant tumors, except skin basal cell carcinoma and cervical carcinoma in situ;
* 4. Accompanied by uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases and other diseases;
* 5. Primary central nervous system lymphoma;
* 6. Left ventricular ejection fraction ≤ 50%;
* 7. Laboratory test values at the time of screening (unless due to lymphoma); A. Neutrophils <1.5*109/L; B. Platelet <75*109/L; C. ALT or AST were 2 times higher than the upper limit of normal, AKP and bilirubin were 1.5 times higher than the upper limit of normal.

D. Creatinine levels higher than 1.5 times the upper limit of normal

* 8. Other concurrent and uncontrolled medical conditions that the investigator believes will affect patient participation in the study.
* 9. Patients with mental illness or other patients known or suspected to be unable to fully comply with the study protocol;
* 10. Pregnant or lactating women;
* 11. People living with HIV.
* 12. Patients with positive HbsAg test results need to undergo HBV DNA test, and can be enrolled before turning negative. In addition, if the HBsAg test result is negative, but the HBcAb test is positive (regardless of the HBsAb status), HBV DNA test should also be performed. If the result is positive, the treatment should also be negative before admission.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS（Progression-free survival） | 1-year
  PFS, defined as the time from treatment to the first occurrence of disease progression or relapse using the 2014 Lugano Response Criteria or death due to any cause, whichever occurs first; as determined by the investigator

SECONDARY OUTCOMES:
CRR（Complete response rate） | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  CR rate at the end of treatment by FDG-PET defined as the proportion of participants with CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator
OS（overall survival） | 2-year
  OS defined as the time from treatment to death from any cause
ORR（overall response rate） | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  ORR at treatment completion or discontinuation defined as the proportion of participants with partial response (PR) or CR at the end of treatment according to the 2014 Lugano Response Criteria; as determined by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- No. 197 Ruijin 2nd Road, Huangpu District, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No